CLINICAL TRIAL: NCT02421237
Title: Randomized Controlled Trial of Treatment for Internalized Stigma in Schizophrenia
Brief Title: Trial of Treatment for Internalized Stigma in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Jay College of Criminal Justice, City University of New York (Other)
Collaborators: Rutgers University (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH094310-02 (NIH)
Record Dates: First submitted 2015-04-10; First posted 2015-04-20 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition (Experimental): Narrative enhancement and cognitive therapy (NECT) groups. Structured psychoeducational and skills-training groups focused on self-stigma and its impact on people with schizophrenia
  Interventions: Behavioral: Narrative Enhancement and Cognitive Therapy
- Control condition (Active Comparator): Supportive group therapy groups. Unstructured supportive groups not focused on self-stigma.
  Interventions: Behavioral: Supportive Group Therapy

INTERVENTIONS:
Behavioral: Narrative Enhancement and Cognitive Therapy
  Arms: Experimental condition
Behavioral: Supportive Group Therapy
  Arms: Control condition

SUMMARY:
The purpose of the present study is to build upon the investigators' previous exploratory intervention development study by conducting an adequately-powered, randomized controlled trial of the Narrative Enhancement/Cognitive Therapy (NECT) intervention among persons with schizophrenia-spectrum disorders.

DETAILED DESCRIPTION:
Internalized (or self) stigma develops when people with mental illness become aware of stigmatizing attitudes held by many in society about mental illness (e.g., dangerousness, incompetence, inability to work), perceive these attitudes as being legitimate, and apply them to themselves. There is substantial evidence that internalized stigma is strongly negatively linked to both the objective (e.g., social functioning) and subjective (e.g., self-esteem and well-being) components of recovery for persons with schizophrenia, and that these effects operate independent of symptom-related disability. Nevertheless, few efforts have been made to develop treatment to address this issue. Previously, the investigators were funded to develop a group-based intervention (R34MH082161) combining cognitive-behavioral therapy and narrative psychotherapy to address internalized stigma among people with severe mental illness. The purpose of the present study is to build upon the investigators' previous exploratory intervention development study by conducting an adequately-powered, randomized controlled trial of the Narrative Enhancement/Cognitive Therapy (NECT) intervention among persons with schizophrenia-spectrum disorders. The investigators will screen 500 persons at two sites (Newark, New Jersey and Indianapolis, IN) for evidence of moderate or elevated internalized stigma. They will conduct a randomized study of NECT versus supportive group therapy in a sample of 175 individuals meeting Structured Clinical Interview criteria for schizophrenia-spectrum disorders. Randomization will be stratified by baseline self-stigma severity (moderate or elevated), to ensure roughly equal numbers of participants for each stratum. Participants will complete baseline, post-treatment, 3-month post treatment and 6-month post treatment assessments of internalized stigma, psychiatric symptoms, insight, self-esteem, hopelessness, coping, narrative coherence and social functioning. The specific aims of the project are: 1) Conduct a randomized study of the effectiveness of NECT, comparing outcomes for 175 persons with schizophrenia-spectrum disorder randomly assigned to NECT or supportive group therapy, 2) Examine the mediating impact of changes in narrative coherence and in the use of problem-centered coping strategies on outcomes for persons assigned to the NECT treatment. The intervention can have important implications for enhancing usual care services to reduce disability for people with schizophrenia, and therefore has potentially important implications for improving the public health.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia-spectrum disorder (schizophrenia or schizoaffective)
* Elevated internalized stigma

Exclusion Criteria:

* Current substance dependence
* Inability to speak English
* Inability to provide informed consent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Internalized Stigma of Mental Illness Scale | Up to 11 months post baseline
Change in Beck Hopelessness Scale | Up to 11 months post baseline
Change in Rosenberg Self-Esteem Scale | Up to 11 months post baseline

SECONDARY OUTCOMES:
Change in Heinrichs Quality of Life Scale | Up to 11 months post baseline

CONTACTS AND LOCATIONS:
Locations (1):
- John Jay College, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No